CLINICAL TRIAL: NCT07144163
Title: A Randomized, Double-Blind, Multicenter, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Atumelnant in Adult Participants With Classic Congenital Adrenal Hyperplasia (Calm-CAH)
Brief Title: A Study to Evaluate Atumelnant in Adults With Congenital Adrenal Hyperplasia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRN04894-12; 2024-519579-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Congenital Adrenal Hyperplasia; Classic Congenital Adrenal Hyperplasia
Keywords: Congenital Adrenal Hyperplasia; CAH; CRN04894; Atumelnant; Adult; Calm-CAH
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Atumelnant tablet, administered orally, once daily for 32 weeks.
  Interventions: Drug: Atumelnant
- Placebo (Placebo Comparator): Matching placebo, administered orally, once daily for 32 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atumelnant — Atumelnant, tablets, once daily by mouth
  Other Names: CRN04894
  Arms: Treatment
Drug: Placebo — Placebo, tablets, once daily by mouth
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, PK, and PD of atumelnant in adults with classic CAH due to 21-OHD.

DETAILED DESCRIPTION:
This is a Phase 3, global, multicenter, randomized, double-blind, placebo-controlled study in adult participants (male or female age ≥18 to <75 years) with classic CAH due to 21-OHD who have been on a stable regimen of GCs for at least 2 months to evaluate efficacy, safety, PK, and PD of atumelnant administered once per day. Following a 3- to 6-week Screening Period, eligible participants will enter the Treatment Period where they will be randomly assigned in a 2:1 ratio to receive either atumelnant 80 mg once daily (with an option for dose escalation to 120 mg once daily at Week 20) or placebo.

A total of approximately 150 participants may be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between ≥18 to <75 years of age at the time of signing the ICF.
2. Willing and able to understand and adhere to the study procedures as specified in the protocol and comply with the study treatment.
3. Have classic CAH due to 21-OHD confirmed by the Investigator and approved by the Medical Monitor.
4. Participants with levels of morning serum A4 as follows:

   * A4 >ULN and treated with <11 mg/m2/day (physiologic) GC doses
   * OR normal A4 (above mid-range to ≤ULN) and treated with ≥15 mg/m2/day GC doses
   * OR A4 >ULN and treated with ≥11 mg/m2/day GC doses.
5. On a stable (defined as no dose change of >5 mg/day hydrocortisone equivalent within 2 months prior to Screening) regimen of GC replacement (e.g., hydrocortisone, prednisolone, prednisone, methylprednisolone, meprednisone, dexamethasone, cortisone acetate) at the time of informed consent.
6. If treated with mineralocorticoids (fludrocortisone), the dose should be stable for at least 2 months prior to Screening without orthostatic hypotension, and with serum sodium and potassium in the normal range.
7. If on estrogen therapy (any route), the dose must be stable for at least 3 months prior to Screening.

Exclusion Criteria:

1. Diagnosis of any form of CAH other than classic 21-OHD.
2. History of bilateral adrenalectomy, hypopituitarism, or other condition requiring chronic GC therapy.
3. Clinically significant medical condition or abnormal laboratory tests, as judged by the Investigator, other than CAH.
4. Concomitant mental condition rendering him/her unable to understand the nature, scope, and possible consequences of the study, and/or evidence of poor compliance with medical instructions.
5. History of cancer excluding cured/treated dermal squamous or basal cell carcinoma or cervical carcinoma in situ.
6. Women who are pregnant or lactating or, if of childbearing potential, who are unwilling to use highly effective contraception as described in this study. Male participants who are unwilling to use highly effective contraception as described in this study.
7. Known history of, or concern for, risk of hypersensitivity reaction to atumelnant or any of its excipients.
8. Participants with an increased risk of developing adrenal insufficiency as judged by the Investigator.
9. Severe erythrocytosis as judged by the Investigator.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with morning post-GC A4 ≤ ULN who are on physiologic GC replacement. | Week 32

SECONDARY OUTCOMES:
Percent change from baseline of morning pre-GC A4 | Week 2
Percent change from baseline of morning pre-GC 17-OHP | Week 32
Proportion of participants with morning pre-GC A4 ≤ ULN who are on physiologic GC replacement | Week 32
Percent change from baseline in GC daily dose when morning post-GC A4 ≤ ULN | Week 32

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Crinetics Study Site, Herston, Queensland
  - Crinetics Study Site, Woolloongabba, Queensland
  - Crinetics Study Site, Adelaide, South Australia
  - Crinetics Study Site, Parkville, Victoria
  - Crinetics Study Site, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No